CLINICAL TRIAL: NCT03519087
Title: Informed Decisions and Patient Outcomes: An Interdisciplinary Approach to Chronic Hip Pain
Brief Title: Nonarthritic Hip Disease Evaluation And Treatment
Acronym: NEAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The planned 15-month recruitment period was completed.
Sponsor: Ohio State University (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie Di Stasi, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017H0340
Record Dates: First submitted 2018-03-27; First posted 2018-05-08 (Actual); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Clinical Decision Making; Nonarthritic Hip Disease
MeSH Terms: interventions — Posture; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Interdisciplinary Evaluation (Experimental): Participants will receive an Interdisciplinary Evaluation for Nonarthritic Hip Disease from a hip arthroscopist, followed by an examination from a physical therapist, and then will participate in a shared decision-making process with both providers to determine a plan of care.
  Interventions: Other: Interdisciplinary Evaluation for Nonarthritic Hip Disease
- Standard Evaluation (No Intervention): Participants will receive a standard-of-care evaluation from a hip arthroscopist who will then determine the plan of care with the participant.
- Posture and Movement Training (Experimental): Participants will receive six training sessions with a physical therapist over a 3-week period.
  Interventions: Other: Posture and Movement Training
- 3-week Wait Period (No Intervention): Participants will undergo a 3-week wait period. They will be instructed to not receive any treatment (e.g. chiropractic services, physical therapy, medication, surgery, injections) for their hip symptoms during this time.
- Observational Arm (Other): Participants who refuse randomization to receive posture and movement training may continue participation in an observational group. These participants complete the same baseline and follow-up testing but proceed with their treatment-of-choice during the 3-week intervention period.
  Interventions: Other: Treatment-of-choice

INTERVENTIONS:
Other: Interdisciplinary Evaluation for Nonarthritic Hip Disease — The hip arthroscopist will conduct his or her standard-care evaluation including subjective interview, patient history, imaging, and physical examination. The physical therapist will conduct an assessment of posture and movement during sitting, standing, squatting, and walking. After providers discuss their findings, they will discuss the plan of care with the participant.
  Arms: Interdisciplinary Evaluation
Other: Posture and Movement Training — Physical therapists will lead participants through an intervention protocol to normalize seated and standing posture and function movement. Verbal, visual, and tactile cues, along with strengthening exercises will be provided to train posture and movement.
  Other Names: Movement Pattern Training
  Arms: Posture and Movement Training
Other: Treatment-of-choice — Participants may proceed with any treatment-of-choice, which may or may not have been recommended by their health care provider(s). Treatments will be recorded, but not controlled.
  Other Names: Standard care
  Arms: Observational Arm

SUMMARY:
The investigators aim to understand how interdisciplinary care influences decisions, expectations, and outcomes for patients with non-arthritic hip disease (NAHD). Patients presenting to the Ohio State University Wexner Medical Center (OSUWMC) Hip Preservation Clinic will be approached for participation. All participants will proceed with their scheduled, standard-care physician evaluation. Participants without NAHD will be excluded. Participants will then be randomized to receive a same-day physical therapist (PT) evaluation. This PT evaluation is not a standard-care practice in the clinic, this was added for research. All participants will complete expectation surveys before and after their evaluation(s). The clinicians will discuss their recommended plan with the patient and the patient will record a final treatment decision and outcome expectations. Participants will then be randomized to either receive posture and movement training (PMT) for 3 weeks or undergo a 3-week wait period. All participants will be required to withhold any treatment during this 3-week period (except PMT in the PMT group). The 3-week wait period for the no-PMT group is aligned with current clinical processes for time from physician evaluation to start of treatment. All participants may proceed with any further interventions (including PMT) after the 3-week period, but none will be provided/required as part of research. Patient-reported outcomes and clinical tests will be recorded before and after the 3-week period, and 3 and 6 months later. Adding a PT evaluation to the physician visit provides no additional risk because the PT evaluation includes similar clinical tests to the physician and movement analysis during tasks participants complete during daily life. Clinical tests before/after the 3-week intervention period may produce muscle soreness that should resolve within 2 days. Understanding how interdisciplinary care influences expectations and outcomes can inform clinicians regarding the effectiveness of interdisciplinary collaboration.

DETAILED DESCRIPTION:
The clinical evaluation by the physician is standard-of-care and performed as part of potential participants' scheduled appointment. Participants in this study will complete a HIPAA authorization to allow data from their clinical evaluation by the physician to be utilized for this study, including any imaging the physician used in their clinical evaluation and the evaluation note entered into the participant's electronic health record. The physician notes are standardized, allowing streamlined data analysis from the electronic health record.

Research activities to occur the same day as the informed consent process include randomization to receive or not receive a clinical evaluation by a physical therapist along with surveys for treatment decisions, expected outcomes, and patient-reported function. A small sub-group of patients will also complete interviews to identify how they felt about their evaluation that day. The HIPAA authorization will also allow the data from the physical therapy evaluation and any subsequent posture and movement training at OSUWMC to be utilized for this study.

Regardless of randomization to receive or not receive a same-day physical therapy evaluation in the physician clinic, all participants will be randomized to receive posture and movement training (PMT) or undergo a 3-week wait period. Participants who are randomized to receive PMT as part of this research study will schedule based on their availability, twice weekly for 3 weeks with an OSUWMC Sports Medicine physical therapist who also hold IRB-approved status as research personnel. Participants will be made aware during the informed consent process that any PMT they receive as part of this study will be their responsibility to pay for using either self-pay or insurance-based methods.

Participants who refuse randomization to receive PMT will be offered to participate in the observational group. These participants proceed with the same baseline and follow-up testing, but continue with their treatment-of-choice rather than an assigned treatment during the 3-week intervention period.

All participants will complete baseline and follow-up biomechanical and clinical follow-up testing in the Motion Analysis and Performance Laboratory. Biomechanical testing involves using 3-dimensional motion capture techniques to analyze movement during 3 functional tasks including walking, sit-to-stand, and a forward tap-down. Clinical testing involves obtaining anthropometric measures, hip strength, patient-reported function, and planned treatment decisions with respective expected outcomes. A small sub-group of patients will also complete interviews at these testing sessions to identify how they feel about the intervention (wait or posture & movement training).

Posture and movement training involves the physical therapist prescribing therapeutic exercises and activities to improve posture and movement (Harris-Hayes 2016), focusing heavily on extrinsic cueing (Benjaminse 2015). Therapeutic exercises and activities will be individualized based on the participant's presentation and will progress according to pain and quality of movement from double-leg to single-leg activities and from functional to more dynamic tasks.

Participants who are randomized to undergo a 3-week wait period will be required to withhold any treatment during the 3-week wait period. These participants will complete the same testing as the participants in the PMT group (see next paragraph). These participants will not receive any intervention during the 3-week wait period; however, after their first follow-up testing session (within 1 week of completing the 3-week wait period), these participants may proceed with any intervention of their choice. The participants in the PMT group may also proceed with any intervention after their first follow-up testing session. These follow-up interventions will not be provided or required as part of the research study, but participants will be asked to report if they completed any follow-up interventions between their first follow-up testing session and their 3month and 6month follow-up testing sessions.

Follow-up testing will occur within 1-week of completing the 3-week intervention period. At this point, participants in both the PMT and no-PMT groups may proceed with any intervention (i.e. surgery, injection, physical therapy). All participants will perform additional follow-up testing at 3- and 6-months post-intervention.

Qualitative interviews will be conducted to evaluate how physicians and physical therapists involved in the study feel about the evaluation and treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old NAHD diagnosis

Exclusion Criteria:

* Osteoporosis or rheumatoid arthritis
* Systemic health condition
* Legal representative required for treatment decisions
* Bilateral symptoms
* Current spine, hip, knee, or ankle surgery or major injury*
* Pregnancy
* Total hip arthroplasty candidate (Tönnis grade > 2)
* Periacetabular osteotomy candidate (lateral center edge angle<20, anterior center edge angle<18, acetabular index >10)

  * Participants with history of spine, hip, knee, or ankle surgery or major injury will be evaluated by the physician to determine appropriateness for evaluation (and treatment) by a physical therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Di Stasi, PhD, PT, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center Jameson Crane Sports Medicine Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
At this time, our IPD will be shared with researchers listed on the funding mechanisms for this project. When submitting manuscripts, IPD will be available upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were excluded from the study before assignment to groups (interdisciplinary vs. standard)
Period: Clinic Evaluation
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Started | 55 | 57 | 0 | 0 | 0
Received Assigned Intervention | 54 | 57 | 0 | 0 | 0
Confirmed Diagnosis by Physician | 39 | 39 | 0 | 0 | 0
Completed | 39 | 39 | 0 | 0 | 0
Not Completed | 16 | 18 | 0 | 0 | 0
Not completed — Physician Decision | 15 | 18 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Period: Re-randomization for Treatment
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Started | 39 | 39 | 0 | 0 | 0
Completed | 12 | 7 | 0 | 0 | 0
Not Completed | 27 | 32 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 29 | 0 | 0 | 0
Not completed — Not appropriate | 2 | 3 | 0 | 0 | 0
Period: Laboratory Testing
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Started | 0 | 0 | 6 (From interdisciplinary (4) or standard (2) evaluation from Period 1) | 6 (From interdisciplinary (4) or standard (2) evaluation from Period 1) | 7 (From interdisciplinary (4) or standard (3) evaluation from Period 1)
Baseline Lab Testing | 0 | 0 | 5 | 4 | 3
Completed | 0 | 0 | 4 | 2 | 1
Not Completed | 0 | 0 | 2 | 4 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The participants who met all eligibility criteria and had non-arthritic hip disease diagnosed by the physician were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 41 (11) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 28 | 30 | 58
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78
Decisional Conflict [Mean (Standard Deviation); unit: units on a scale] — Decisional conflict was measured using the Decisional Conflict Scale ranging from 0 (no conflict, better outcome) to 100 (high conflict, worse outcome).
  units on a scale | 35.0 (19.6) | 40.1 (18.6) | 37.6 (19.2)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Plan
Description: Participants will indicate their planned treatment(s)
Time Frame: Post-evaluation, same-day (approximately 5-10min after evaluation)
Population: Participants from Period 1 (Clinic evaluation) were analyzed for this primary outcome measure based on interdisciplinary or standard evaluation. This outcome measure was not a planned outcome for Period 3 (Laboratory testing) and thus, values are not reported for posture and movement training, 3-week wait period, or observational groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Number analyzed (Participants) | 39 | 39 | 0 | 0 | 0
Participants
  Physical Therapy included in treatment plan | 26 | 19 |  |  |
  Surgery included in treatment plan | 19 | 19 |  |  |
  Injection included in treatment plan | 13 | 21 |  |  |

2. Primary Outcome: Decisional Conflict
Description: Participants will report decisional conflict related to their treatment plan. Decisional conflict was measured using the Decisional Conflict Scale ranging from 0 (no conflict, better outcome) to 100 (high conflict, worse outcome).
Time Frame: Pre-evaluation, 10min Post-evaluation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Number analyzed (Participants) | 39 | 39 | 0 | 0 | 0
units on a scale
  Pre-evaluation decisional conflict | 35.0 (19.6) | 40.1 (18.6) |  |  |
  Post-evaluation decisional conflict | 10.2 (11.2) | 16.5 (13.6) |  |  |

3. Secondary Outcome: Themes From Provider Interviews
Description: Qualitative interviews will be conducted with study providers both before patient participant enrollment and after study completion to collect information on how they feel about the evaluation protocols. Qualitative analysis of this data will count responses based on themes. Data for this report will be provided as the total number of responses (across all providers) that fell within each theme at both time points. Each provider could provide multiple responses.
Time Frame: Pre-enrollment (2-7days before patient participant recruitment began), Post-enrollment (1-7 days after patient participant recruitment ended)
Population: The orthopaedic surgeons (n=2) and one physical therapist (n=1) from the study were interviewed and number of responses during the interviews were totaled based on theme. Each provider could have multiple responses. These providers are not associated with a specific arm or group of patient participants.
Measure: Number; unit: number of responses for each theme
Groups:
- Pre-enrollment; Post-enrollment: The orthopaedic surgeons (2) and physical therapist (1) who participated as study clinicians were interviewed regarding their opinions of the interdisciplinary evaluation.
Arm/Group | Pre-enrollment | Post-enrollment
Number analyzed (Participants) | 3 | 3
number of responses for each theme
  Implementation | 11 | 13
  Interdisciplinary Evaluation | 10 | 13
  Time | 6 | 8
  Patient Response | 12 | 11
  Clinical Reasoning | 7 | 9
  Environment | 2 | 5

4. Secondary Outcome: Participant Protocol Opinions
Description: Participants will be interviewed to collect information on how they feel about the 1) evaluation protocol(s) and 2) treatment/wait period protocols.
Time Frame: 20min post-evaluation, 4 weeks post-evaluation
Population: Data were not collected.
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation | Posture and Movement Training | 3-week Wait Period | Observational Arm
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Decisional Conflict
Description: Participants will report decisional conflict related to their treatment plan. Decisional conflict was measured using the Decisional Conflict Scale ranging from 0 (no conflict, better outcome) to 100 (high conflict, worse outcome). Baseline scores for participants in Period 3 (Laboratory testing) were obtained from participants' post-evaluation surveys from Period 1 (clinic evaluation).
Time Frame: 10min post-evaluation, 4-week laboratory visit
Population: Participants from Period 3 (Laboratory testing) were analyzed for this secondary outcome measure based on treatment group (Posture & movement training, wait period, or observational). This outcome measure was not a planned follow-up outcome for Period 1 (Clinic evaluation) and thus, values are not reported for interdisciplinary and standard groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posture and Movement Training | 3-week Wait Period | Observational Arm | Interdisciplinary Evaluation | Standard Evaluation
Number analyzed (Participants) | 4 | 2 | 1 | 0 | 0
units on a scale
  Post-evaluation decisional conflict | 13.2 (10.3) | 14.8 (20.9) | 0 (0) |  |
  4-week decisional conflict | 14.0 (16.2) | 13.2 (9.9) | 0.0 (0.0) |  |

6. Secondary Outcome: Patient-reported Hip Function
Description: Participants will complete validated, reliable surveys for hip function (the Hip Outcome Score Activities of Daily Living [HOSADL] was used and is scored from 0-100 with 0 representing the worst function and 100 representing the best function). Baseline scores for participants in Period 3 (Laboratory testing) were obtained from participants' post-evaluation surveys from Period 1 (clinic evaluation).
Time Frame: 10min post-evaluation, 4-week laboratory visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Posture and Movement Training | 3-week Wait Period | Observational Arm | Interdisciplinary Evaluation | Standard Evaluation
Number analyzed (Participants) | 4 | 2 | 1 | 0 | 0
units on a scale
  Post-evaluation HOSADL | 52.9 (21.7) | 72.6 (29.8) | 89.0 (0) |  |
  4-week HOSADL | 68.2 (20.0) | 77.2 (25.9) | 92.6 (0) |  |

7. Secondary Outcome: Movement Mechanics
Description: 3-dimensional movement mechanics will be collected during functional tasks including walking and rising from a chair
Time Frame: Baseline laboratory visit, 4-week laboratory visit
Population: Movement mechanics were not a planned variable for Period 1 (Clinic evaluation), but were a planned secondary variable for Period 3 (Laboratory testing). Collected data for the 7 participants who completed 4-week testing required extensive processing and resources that were not available due to loss of funding and personnel.
Arm/Group | Posture and Movement Training | 3-week Wait Period | Observational Arm | Interdisciplinary Evaluation | Standard Evaluation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Decisional Regret
Description: Participants will report decision regret related to their treatment plans
Time Frame: Day of enrollment, after all evaluations are complete
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Decisional Regret
Description: Participants will report decision regret related to their treatment plans
Time Frame: 4 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Hip Strength
Description: Strength of hip abductors, adductors, flexors, extenders, internal and external rotators will be collected during maximal voluntary isometric contractions
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the 15-month recruitment period and up to the 4-week follow-up for any participants who underwent treatment as part of the trial.
Description: Adverse events were defined per the clinicaltrials.gov definitions. Adverse events that were (1) reported by participants to study personnel or study clinicians or (2) identified by study personnel or study clinicians were recorded.
Arm/Group | Interdisciplinary Evaluation | Standard Evaluation
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

LIMITATIONS AND CAVEATS:
Seventy-eight (78) participants were included from the 15-month recruitment period (81% of the target n=96). Randomization for interdisciplinary vs. standard evaluation had to occur before physician evaluation, modified from the original protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03519087/Prot_003.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03519087/SAP_004.pdf
  • Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03519087/ICF_005.pdf